CLINICAL TRIAL: NCT01077635
Title: An Observational Multi-cohort Study on the Use of Fosamprenavir-Ritonavir Among HIV-infected Children and Adolescents in Europe
Brief Title: PENTA Fosamprenavir Study
Status: Completed | Type: Observational
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 112880
Record Dates: First submitted 2010-02-25; First posted 2010-03-01 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2012-01

CONDITIONS: Infection, Human Immunodeficiency Virus
Keywords: HIV; Antiretroviral therapy; protease inbitor; fosamprenavir; paediatrics
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — BID protein, human; Ritonavir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HIV-1 infected children aged 6 ≤ 18 years: HIV-1 infected children aged 6 ≤ 18 years currently or having ever been exposed to FPV/RTV; this is the indicated group for the licensed dose in the paediatric population.
  Interventions: Drug: Exposure to licensed dose of FPV (+/- 20% of 18mg/kg BID + RTV)

INTERVENTIONS:
Drug: Exposure to licensed dose of FPV (+/- 20% of 18mg/kg BID + RTV) — HIV-1 infected children currently or having ever been exposed to FPV (+/- 20% of 18mg/kg BID + RTV)

SUMMARY:
Twice daily fosamprenavir, in combination with low dose ritonavir (FPV/RTV BID), is indicated for the treatment of HIV-infected adults, adolescents and children of 6 years of age and above for use in combination with other anti-HIV medicines. Safety data from two GlaxoSmithKline (GSK) clinical trials (APV29005 - involving twice-daily doses of FPV with or without RTV and APV20003 - with once daily dosing of FPV/RTV among 2-18 year olds) indicated that gastrointestinal events were the most commonly reported AEs, but that the majority of events were mild and of short duration. Treatment emergent grade 3 / 4 neutropenia was reported in 20% of children in the APV20003 trial; and neutropenia was identified as a potential safety concern by the European Medicines Agency (EMEA). The objectives of this study were to conduct an observational cohort study of the usage and safety of FPV/RTV in children and adolescents (aged 6 ≤ 18 years) with HIV infection in several European HIV paediatric cohorts. Data will be collected for 3 years (2008, 2009 and 2010).

DETAILED DESCRIPTION:
ViiV Healthcare is the new sponsor of this study, and GlaxoSmithKline is in the process of updating systems to reflect the change in sponsorship.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected children aged 6-18 years exposed to licensed paediatric dose of FPV/RTV January 1 2008 (or date of exposure to FPV if earlier to this but still exposed at 1/1/2008) from the participating cohorts

Exclusion Criteria:

-

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Seven paediatric HIV cohorts participating in the European Pregnancy and Paediatric HIV Cohort Collaboration (EPPICC) as follows: French Perinatal Cohort Study / Enquête Périnatale Français; Hospital St.Pierre Cohort, Brussels; Italian Register for HIV-infection in Children; Madrid Cohort of HIV-infected Children; Spanish Perinatal Cohort Study [NENEXP], Catalonia, Spain; UK National Study of HIV in Pregnancy and Childhood [NSHPC] & Collaborative HIV Paediatric Study [CHIPS]; and the "Victor Babes" Hospital Cohort, Romania.
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2008-10; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Number of children on licensed dose of FPV/RTV | Assessed at 1, 2 and 3 years post exposure

SECONDARY OUTCOMES:
Reason for stopping FPV | Assessed at 1, 2 and 3 years post exposure
Laboratory tests for absolute neutrophil counts (ANC), lipids (total cholesterol [TC] and triglycerides [TG]), and alanine transaminase (ALT) | Assessed at 1, 2 and 3 years post exposure

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare